CLINICAL TRIAL: NCT00777738
Title: A Phase IIA Trial Testing the Efficacy of Bortezomib (Velcade(R)) in Patients With Advanced Waldenström Macroglobulinemia
Brief Title: Efficacy of Bortezomib (Velcade(R)) in Patients With Advanced Waldenström Macroglobulinemia
Acronym: WM2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P060207
Record Dates: First submitted 2008-10-16; First posted 2008-10-22 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2008-10

CONDITIONS: Waldenstrom Macroglobulinemia
Keywords: Advanced Waldenström's macroglobulinemia; Bortezomib; Dexamethasone; Safety; Efficacy
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bortezomib (Experimental): bortezomib
  Interventions: Drug: BORTEZOMIB

INTERVENTIONS:
Drug: BORTEZOMIB — * Bortezomib (Velcade(R)): 1.3 mg/m2 on Days 1, 4, 8, and 11 every 21 days for 2 cycles (IV route, push).
  * For responding patients : up to 6 cycles
  * For non responding patient : Adjunction of dexamethasone (HD DXM) : 20 mg Days 1,D2, D 4,D 5, D8, D9 and D 11,D12 every 21 days

SUMMARY:
This trial is designed to evaluate the efficacy and toxicity of Bortezomib , an inhibitor of proteasome used in multiple myeloma, in patients with advanced Waldenström's Macroglobulinemia disease.

DETAILED DESCRIPTION:
Open, prospective, multicenter, non controlled phase IIA trial

Primary objectives Evaluation of the efficacy and safety of Velcade in monotherapy for patients with advanced stage Waldenström Macroglobulinemia.

Secondary objectives Evaluation of the activity of the association of High Dose Dexamethasone (HD DXM) with Velcade for patients resistant to Velcade Alone For all patients

* Overall survival
* Safety
* Quality of life
* Duration of response

sample size: With type I error alpha of 5% and type II error beta of 20% and a two-sided test, the number of patients needed in this study is 34 Number of centers: 28 Centers participating to the French cooperative group CLL/WM

ELIGIBILITY:
Inclusion Criteria:

● Established diagnosis of Waldenström macroglobulinemia (the 2nd Workshop on Waldenstrom's macroglobulinemia)

Patient must have had 1 (or 2) lines of chemotherapy containing alkylating agent and/or Fludarabine :and /or monoclonal antibody and must have :

* Life expectancy > 3 months
* Age > 18 years
* ECOG performance status 0-1-2
* ANC > 1 x 109/L
* Creatinine clearance, calculated according to the formula of cockcroft and Gault > 40 ml/min
* Total bilirubin < 2x ULN
* ASAT, ALAT < 2x ULN
* A negative serum pregnancy test one week prior to treatment must be available both for pre-menopausal women and for women who are < 2 years after the onset of menopause
* Adequate contraceptive methods for males and pre-menopausal females for 6 months after treatment discontinuation.
* Written informed consent
* Platelets> 100X 109

Exclusion Criteria:

* Active secondary malignancy or chemotherapy/radiotherapy for any neoplastic disease other than Waldenström macroglobulinemia prior to the study
* Medical condition requiring the long-term (estimated to be more than one month) use of oral corticosteroids
* Patients with active bacterial, viral or fungal infection
* Known infection with HIV, Hepatitis B (except post vaccinal profile) or C
* Treatment with any, other investigational agent or participating in another trial within 30 days prior to entering this study
* Lactation/pregnancy
* Concurrent severe diseases which exclude the administration of therapy heart insufficiency NYHA grade III/IV, LEVF < 50% and or RF < 30%, myocardial infarction within the past 6 months prior to study
* Severe pulmonary or heart problems (acute diffuse pulmonary and pericardial disease)
* Severe chronic obstructive lung disease with hypoxemia
* Severe diabetes mellitus
* Hypertension difficult to control
* Impaired renal function with creatinine clearance < 40 ml/min according to the formula of Cockcroft and Gault
* Cerebral dysfunction
* Richter's syndrome
* Neuropathy> grade 1
* Positive Beta HCG
* Severe Hepato cellular alteration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Complete and partial remission, defined by the 2nd Workshop on Waldenstrom's macroglobulinemia | 3 months and 6 months

SECONDARY OUTCOMES:
Duration of the response | during the study
Overall survival | during the study
Quality of life | months 0, 3, 12, 24

CONTACTS AND LOCATIONS:
Overall Officials: Véronique LEBLOND, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital La Pitie Salpetriere, Paris, France